CLINICAL TRIAL: NCT02259868
Title: Randomized Single Dose Multiple Crossover Relative Bioavailability Trial of New Tablet Formulations and Suspension Formulation Compared to Current (1B) Formulation of BILR 355 BS in Healthy Male Volunteer Subjects
Brief Title: Study of New Tablet Formulations and Suspension Formulation Compared to Current (1B) Formulation of BILR 355 BS in Healthy Male Volunteer Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1188.5
Record Dates: First submitted 2014-10-07; First posted 2014-10-09 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Healthy
MeSH Terms: interventions — Dosage Forms; Sodium Dodecyl Sulfate; Ritonavir

ARMS (4):
- Group A (Experimental): randomized sequence of current low dose formulation (3 tablets) and high dose (1 tablet) BILR 355 BS 1B formulation, separated by 14-day washout
  Interventions: Drug: BILR 355 BS /1B, current low dose formulation; Drug: BILR 355 BS /1B, current high dose formulation; Drug: Ritonavir
- Group B (Experimental): randomized sequence of BILR 355 BS (JM) + SDS formulation low dose (2 tablets) ,BILR 355 BS (HM) + SDS formulation low dose (2 tablets), BILR 355 BS high dose 1B formulation (4 low dose tablets), separated by 14-day washout
  Interventions: Drug: BILR 355 BS /1B, current low dose formulation; Drug: BILR 355 BS - Jet Milled (JM) + Sodium Dodecyl Sulfate (SDS) formulation; Drug: BILR 355 BS - Hammer Milled (HM) + Sodium Dodecyl Sulfate (SDS) formulation; Drug: Ritonavir
- Group C (Experimental): randomized sequence of BILR 355 BS (JM) + SDS formulation high dose (4 tablets) , BILR 355 BS (JM) + SDS formulation mid dose (3 tablets), BILR 355 BS (HM) + SDS formulation high dose (4 tablets), separated by 14-day washout
  Interventions: Drug: BILR 355 BS - Jet Milled (JM) + Sodium Dodecyl Sulfate (SDS) formulation; Drug: BILR 355 BS - Hammer Milled (HM) + Sodium Dodecyl Sulfate (SDS) formulation; Drug: Ritonavir
- Group D (Experimental): randomized sequence of BILR 355 BS Suspension high dose, BILR 355 BS Suspension low dose, current low dose BILR 355 BS 1B formulation (3 tablets) separated by 14-day washout
  Interventions: Drug: BILR 355 BS /1B, current low dose formulation; Drug: BILR 355 BS - Suspension low dose; Drug: BILR 355 BS - Suspension high dose; Drug: Ritonavir

INTERVENTIONS:
Drug: BILR 355 BS /1B, current low dose formulation
  Arms: Group A; Group B; Group D
Drug: BILR 355 BS /1B, current high dose formulation
  Arms: Group A
Drug: BILR 355 BS - Jet Milled (JM) + Sodium Dodecyl Sulfate (SDS) formulation
  Arms: Group B; Group C
Drug: BILR 355 BS - Hammer Milled (HM) + Sodium Dodecyl Sulfate (SDS) formulation
  Arms: Group B; Group C
Drug: BILR 355 BS - Suspension low dose
  Arms: Group D
Drug: BILR 355 BS - Suspension high dose
  Arms: Group D
Drug: Ritonavir

SUMMARY:
1. To investigate the relative bioavailability (BA) of improved tablet formulation candidates to determine which formulation will be developed for use in late Phase II and Phase III clinical trials
2. To investigate the relative BA of the pediatric suspension, compared to the current 1B formulation
3. To investigate the bioequivalence (BE) of BILR 355 BS in two tablet strengths; three 25mg tablets vs. one 75 mg tablet, current 1B formulation

ELIGIBILITY:
Inclusion Criteria:

1. Healthy HIV negative adult male volunteers
2. Age ≥18 and ≤ 60 years
3. BMI ≥18.5 and BMI ≤29.9 kg/m2
4. Ability to give signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local regulations

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Surgery of gastrointestinal tract (except appendectomy)
3. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
4. History of relevant orthostatic hypotension, fainting spells or blackouts
5. Chronic or relevant acute infections
6. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
7. Intake of drugs with a long half-life (>24 hours) within at least one month prior to study drug administration and during the trial
8. Use of drugs within 10 days prior to administration or during the trial which might reasonably influence the results of the trial
9. Participation in another trial with an investigational drug within two months prior to administration or during the trial
10. Current smoker
11. Alcohol abuse (more than 60 g/day)
12. Drug abuse (positive urine test for illicit prescription or non-prescription drugs or drugs of abuse).
13. Blood donation (more than 100 mL within four weeks prior to study drug administration or during the trial)
14. Excessive physical activities (within one week prior to study drug administration or during the trial)
15. Any laboratory value outside the reference range that is of clinical relevance at screening, according to the judgment of the investigator
16. Inability to comply with dietary regimen required by the protocol
17. Infected with hepatitis B or hepatitis C viruses (defined as either being hepatitis B surface antigen, or hepatitis C antibody positive

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2005-06; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Up to 96 hours after drug administration
Cmax (maximum measured concentration of analyte in plasma) | Up to 96 hours after drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | Up to 96 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | Up to 96 hours after drug administration
λz (terminal rate constant in plasma) | Up to 96 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | Up to 96 hours after drug administration
MRTpo (mean residence time of the analyte in the body after po administration) | Up to 96 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | Up to 96 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | Up to 96 hours after drug administration
Number of participants with clinically significant changes in vital signs | Up to day 43 after first drug administration
Number of participants with abnormal changes in clinical laboratory parameters | Up to day 43 after first drug administration
Number of participants with Adverse Events | Up to day 43 after first drug administration